CLINICAL TRIAL: NCT04340596
Title: A Phase I Clinical Trial of the Safety, Tolerability, and Efficacy of IL-15 Superagonist (N-803) With and Without Combination Broadly Neutralizing Antibodies to Induce HIV-1 Control During Analytic Treatment Interruption
Brief Title: Safety, Tolerability, and Efficacy of IL-15 Superagonist (N-803) With and Without Combination Broadly Neutralizing Antibodies to Induce HIV-1 Control During Analytic Treatment Interruption
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Rockefeller University (Other); ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5386; 38639 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2020-03-23; First posted 2020-04-09 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: N-803 only (Experimental): Participants will receive N-803 6 mcg/kg 1 week after Step 2 entry and then every 3 weeks for a total of eight doses.
  Interventions: Biological: N-803 (IL-15 Superagonist)
- Arm B: N-803 in combination with 10-1074 and VRC07-523LS (Experimental): Participants will receive N-803 in combination with 10-1074 and VRC07-523LS as follows:
  * At Step 2 entry:
    * VRC07-523LS 20 mg/kg
    * 10-1074 30 mg/kg
  * At Step 2, week 1: N-803 6 mcg/kg every 3 weeks for eight doses
  * At Step 2, week 9: 10-1074 30 mg/kg
  Interventions: Biological: N-803 (IL-15 Superagonist); Biological: VRC07-523LS; Biological: 10-1074

INTERVENTIONS:
Biological: N-803 (IL-15 Superagonist) — Administered by subcutaneous (SQ) injection
Biological: VRC07-523LS — Administered by intravenous (IV) infusion
  Arms: Arm B: N-803 in combination with 10-1074 and VRC07-523LS
Biological: 10-1074 — Administered by intravenous (IV) infusion
  Arms: Arm B: N-803 in combination with 10-1074 and VRC07-523LS

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of N-803, an IL-15 superagonist, with or without combination broadly neutralizing antibodies (bNAbs), to induce HIV-1 control during analytic treatment interruption (ATI).

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, and efficacy of N-803, an IL-15 superagonist, with or without combination broadly neutralizing antibodies (bNAbs), to induce HIV-1 control during analytic treatment interruption (ATI).

Participants will be screened for eligibility and undergo leukapheresis, and a subset will also undergo optional rectal biopsy and/or lymph node fine needle aspirations (FNAs) (Step 1).

After pre-entry and determination of eligibility in Step 1, participants will be randomized before Step 2 entry to either the N-803 only arm (Arm A) or the N-803 with combination bNAbs arm (Arm B):

* Arm A will receive a dose of N-803, 6 mcg/kg, subcutaneously 1 week after Step 2 entry and then every 3 weeks for a total of eight doses (during the first 22 weeks).
* Arm B will receive the following (during the first 22 weeks):

  * Combination bNAb at Step 2 entry with VRC07-523LS dosed at 20 mg/kg and 10-1074 dosed at 30 mg/kg, intravenously;
  * A dose of N-803, 6 mcg/kg, subcutaneously 1 week after Step 2 entry and then every 3 weeks for a total of eight doses;
  * A second dose of 10-1074 at week 9 of Step 2 dosed at 30 mg/kg, intravenously

After completing randomized treatment (Step 2), participants will interrupt antiretroviral therapy (ART) (Step 3) and will be followed closely to monitor for indications for reinitiation of ART (Step 4).

After Step 2 entry, most participants will be followed for approximately 100 weeks across the remaining three study steps (i.e., Steps 2, 3, and 4).

Step 1 will last up to 90 days, Step 2 will last approximately 52 weeks (study intervention), Step 3 will last up to 24 weeks (ATI), and Step 4 will last 24 weeks (ART restart).

ELIGIBILITY:
Inclusion Criteria

* HIV-1 infection
* On ART for at least 96 weeks prior to randomization
* On ART regimen containing an integrase inhibitor and two nucleoside reverse transcriptase inhibitors (NRTIs) or dolutegravir/lamivudine for at least 6 weeks prior to randomization.
* CD4 cell count >450 cells/mm^3 within 90 days prior to randomization
* CD4 cell count nadir ≥200 cells/mm^3.
* Plasma HIV-1 RNA levels of <50 copies/mL for at least 96 weeks prior to randomization
* Select laboratory results within 90 days of randomization
* IC90 to 10-1074 of ≤1.5 mcg/mL, 10-1074 maximum percent inhibition (MPI) ≥98%, and IC80 to VRC07-523LS of ≤1 mcg/mL on the Monogram PhenoSense assay.
* QTcF interval ≤440 msec within 90 days prior to randomization.
* For cisgender women and transgender men of reproductive potential, negative urine or serum pregnancy test within 30 days prior to randomization
* Cisgender women and transgender men of reproductive potential must agree to use two methods of contraception, if participating in sexual activity that could lead to pregnancy.
* Cisgender men and transgender women participants engaging in sexual activity that could lead to pregnancy and who are of reproductive potential must agree to use a barrier method of contraception
* Willingness to abstain from sexual intercourse or use a barrier method of contraception consistently
* Willingness to participate in an ATI.
* Weight >50 kg and <115 kg.
* Completion of pre-entry leukapheresis

Exclusion Criteria

* History of AIDS-defining illness, with the exception of recurrent pneumonia.
* History of or current clinical cardiovascular disease
* Current clinically significant acute or chronic medical condition
* History of HIV-associated neurocognitive disease
* History of an HIV-associated malignancy
* ART initiated during acute HIV infection
* Current receipt of ART other than NRTI and integrase inhibitor.
* Resistance to one or more drugs in two or more ARV drug classes.
* Receipt of any therapeutic HIV vaccine or monoclonal antibody therapy (anti-HIV or otherwise) at any time in the past.
* History of prior immunoglobulin (IgG) therapy.
* History of use of any immunomodulatory medications within 6 months prior to randomization
* Participation in another clinical study of an investigational product currently or within past 12 weeks
* Breastfeeding or pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a Grade ≥3 adverse event (AE) that is at least possibly related to N-803, as judged by the Clinical Management Committee (CMC) | Step 2 week 1 to week 52
Number of N-803 doses completed | From step 2 week 1 to step 2 week 22
  Eight doses of N-803 are scheduled at the distinct time points listed in Time Frame. At each timepoint, dose completion status is recorded. Number of N-803 doses completed is the total number completed doses across all 8 timepoints.
Proportion of participants requiring dose reduction | From step 2 week 4 to step 2 week 22
  Eight doses of N-803 are scheduled at distinct time points (Step 2 weeks 1, 4, 7, 10, 13, 16, 19 and 22). Proportion of participants requiring dose reduction is calculated as the number of participants who receive a reduced dose of N-803 at any of the 7 scheduled doses occurring after the first dose, divided by the total number of participants receiving N-803.
Proportion of participants with plasma HIV-1 RNA <200 copies/mL 8 weeks after interruption of ART | At step 3 week 8

SECONDARY OUTCOMES:
Occurrence of a Grade ≥2 AE without regard to relationship to study treatment | Study entry to participant's last study visit, at approx. study week 100
Occurrence of a Grade ≥2 AE that is at least possibly related to N-803, as judged by the CMC | Step 2 week 1 to week 52
Occurrence of a Grade ≥2 AE that is at least possibly related to VRC07-523LS or 10-1074 | Step 2 week 0 to week 52
Cell-associated HIV-1 RNA | At Step 2 weeks 0, 1, 7, 13, 19, 22, 26 and 32
Measurement of HIV-1 reservoir (dQVOA) | At Step 2 weeks 0, 1, 7, 13, 19, 22, 26 and 32
Measurement of plasma viremia by HIV-1 single copy assay | At step 1 pre-entry evaluation and step 2 weeks 0, 1, 7, 13, 22 and 32
Measurement of intact proviral DNA | At Step 2 weeks 0, 1, 7, 13, 19, 22, 26 and 32
Total HIV-1 DNA | At Step 2 weeks 0, 1, 7, 13, 19, 22, 26 and 32
Proportion of participants with plasma HIV-1 RNA <200 copies/mL at 4, 12 and 24 weeks after interruption of ART in Step 3 | At step 3 weeks 4, 12, and 24
PK parameters: AUC0-τ of 10-1074 | At step 2 weeks 0, 1, 4, 7, 9, 10, 13, 16, 19, 22, 26, 32 and 46
PK parameters: AUC0-τ of VRC07-523LS | At step 2 weeks 0, 1, 4, 7, 9, 10, 13, 16, 19, 22, 26, 32 and 46
Proportion of participants with antidrug antibodies | At step 2 weeks 0, 1, 4, 7, 9, 10, 13, 16, 19, 22, 26, 32 and 46
  Presence of anti-N803, anti-10-1074, and anti-VRC07-523LS antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Wilkin, MD, MPH, Study Chair — Weill Medical College of Cornell University
Locations (14):
- United States (14):
  - Alabama CRS (Site ID# 31788), Birmingham, Alabama
  - UCLA CARE Center CRS, Los Angeles, California
  - UCSD Antiviral Research Center CRS (Site ID: 701), San Diego, California
  - University of California, San Fransisco HIV/AIDS CRS, San Francisco, California
  - Whitman-Walker Institute, Inc. CRS (Site ID: 31791), Washington D.C., District of Columbia
  - Northwestern University CRS, Chicago, Illinois
  - Massachusetts General Hospital CRS (MGH CRS) (Site ID: 101), Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - New Jersey Medical School Clinical Research Center CRS [Site ID: 31786], Newark, New Jersey
  - Columbia P&S CRS, New York, New York
  - Weill Cornell Uptown CRS (Site ID: 7803), New York, New York
  - Chapel Hill CRS (Site ID: 3201), Chapel Hill, North Carolina
  - Case Clinical Research Site, Cleveland, Ohio
  - Penn Therapeutics, CRS (Site ID: 6201), Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://actgnetwork.org/about-actg/templates-and-forms. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.

REFERENCES:
- See also: Related Info — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Related Info — https://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids